Elec**T**rical **I**mpedance **T**omog**R**aphy vs dynamic compli**AN**ce guided positive end-expiratory pressure **T**itration during laparoscopic gynaecological surgery: A multi-centre, prospective randomized trial – **TITRANT Trial** 

## **INFORMED CONSENT FORM**

Approval Number: BM/8893-3/2025

Last updated on March 12, 2025

## **Informed Consent Form**

| December 1 de utification Datas |
|---|
| Research Identification Data: |
| Title of the study: |
| Elec <b>T</b> rical <b>I</b> mpedance <b>T</b> omog <b>R</b> aphy vs dynamic compli <b>AN</b> ce guided positive end-<br>expiratory pressure <b>T</b> itration during laparoscopic gynaecological surgery: A multi-<br>centre, prospective randomized trial – <b>TITRANT Trial</b> |
| Study ID number: |
| BM/8893-3/2025 |
| Location of the study: |
| Principal Investigator: |
| Dr. Zoltán Ruszkai, PhD |
| Head of Department of Anaesthesiology and Intensive Therapy |
| ruszkai.zoltan@florhosp.hu |
| +36-20-915-1978 |
| Participant Data: |
| Name: |
| Mother's name: |
| Place and date of birth: |
| Social Security Number (TAJ): |
| Address: |
| In case of a participant with limited or no legal capacity, the data of the legal representative providing consent: |
| Name: |
| Mother's name: |
| Place and date of birth: |
| Social Security Number (TAJ): |
| Address: |

## Details of the person providing information:

Name:

Position, job title:

Participation in the study is voluntary and completely free from any influence. Consent may be withdrawn at any time, verbally or in writing, without explanation. Withdrawal of consent will not cause any disadvantage for the participant. Should you have any questions, please do not hesitate to ask your attending physician or the investigator leading the study.

Only sign this Consent Form if you have had the opportunity to ask your questions and have received satisfactory answers to all of them.

By signing this Consent Form, you indicate that you voluntarily and without influence agree to participate in the study.

This Consent Form may be withdrawn verbally or in writing at any time, without explanation, and you are free to withdraw from the study at any time.

I declare (in the case of a participant with limited or no legal capacity, we declare together with the legal representative) that:

- I have received both oral and written information:
- I understand the risks and benefits of participating in the study;
- I had the opportunity to ask my questions, and I received satisfactory answers;
- I have given my consent to participate in the study voluntarily and without influence, after receiving prior information;
- I understand that my consent may be withdrawn at any time, verbally or in writing, without explanation;
- I understand that I will be informed of any information that may affect my decision to continue participation in the study;

- I understand that, upon signing, I will receive one original copy each of the information sheet and the consent form;
- I understand that my consent to participate in this study does not nullify my
  rights guaranteed by law, which I may exercise if those involved in conducting
  the study commit negligence or any other error with legal consequences;
- I am aware that I am protected by the relevant data protection laws, and I
  understand that my personal data arising from the study will only be shared in
  compliance with the specific rules laid down in these laws.

| Kistarcsa, 202 month day | |
|---|---|
| Signature of information provider | Signature of participant |
| If the participant or the legal representative cannot read, the valid consent form requires the presence and signatures of two witnesses. | |
| We, the undersigned witnesses, confirm with our signatures that the person intended to be enrolled in the study, or their legal representative, received all possible information, and that the individual and/or their legal representative gave consent to participate voluntarily and free of influence. | |
| Kistarcsa, 202 month day | |
| Signature of information provider | Signature of legal representative |
| Witness 1 | Witness 2 |
| Name: | Name: |
| Address: | Address: |
| ID number: | ID number: |